CLINICAL TRIAL: NCT01376986
Title: Activation of Young Men - Population-Based Randomised Controlled Trial
Acronym: MOPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu Deaconess Institute (Other); City of Oulu (Unknown); Finnish Defense Forces (Other Government); Virpiniemi Sports Institute (Unknown)
Responsible Party: Principal Investigator, Raija Korpelainen, professor, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OKM/98/627/2010
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Obesity; Well-being; Quality of Life; Depression
MeSH Terms: conditions — Obesity; Depression | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Activation (Experimental): All those determined fit for service or who are granted postponement will be included in the activation intervention. The physical activation intervention will be implemented between the call-up and start of military service. The activation group utilises an ICT platform that will be developed.
  Interventions: Behavioral: physical, psychological and social activation
- control (No Intervention): no access to the activation platform

INTERVENTIONS:
Behavioral: physical, psychological and social activation
  Arms: Activation

SUMMARY:
The aim of the study is to investigate different novel IC technologies for promoting physical activity and health and preventing obesity in young men. The purpose is to provide new evidence-based knowledge on the effectiveness of an ICT-based physical activation and to identify factors predicting a positive response.

Specific objectives

* to identify the factors associated with physical activity and physical activity relationship in young men
* to develop an interactive method, based on peer networks, aimed at activating young men with use of their own skills, participation and modern ICT
* to assess the effectiveness of the chosen activation on the physical activity, weight, fitness, health, and relationship towards physical activity among young men

The study population consists of all conscription aged men in the Oulu area in 2011-2013 (n=4000). Conscription-aged men provide a large, population based representative sample of young men. In Finland military service is mandatory and annually all 18-year old men are called for military service. In the call-ups fitness for service is determined based on medical examination.

All those who are determined fit for service or who are granted postponement due to obesity will be invited for the activation intervention study. Those with severe obesity are exempted from service, but will also participate in the trial. After the call-up, the men will be randomised to an intervention group and a control group. The primary outcome variable is change in physical activity.

The study will be conducted during 2011-2015. The study includes technology development (ICT platform), collection of cross-sectional data at the call-ups, and a 6-month physical activity intervention (a randomized controlled trial) implemented between the call-up and start of military service. Game mechanics are integrated into the ICT platform to increase user engagement and participation.

Physical activity, fitness (aerobic and muscular), body composition,lifestyle and psychological and physical health will be followed. In addition, the subjects' entry into military service and its course will be followed.

ELIGIBILITY:
Inclusion Criteria:

* All men born 1995 liable for military service and attending call-ups in Oulu area at 2013

Exclusion Criteria:

* Severe physical or mental illness

Ages: 17 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 507 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
physical activity | 6 months
  physical activity measured continuously over the 6-month trial

SECONDARY OUTCOMES:
weight | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Timo Jämsä, PhD, Study Director — University of Oulu; Matti Mäntysaari, MD, Study Director — Finnish Defense Forces; Raija Korpelainen, PhD, Study Director — raija.korpelainen@odl.fi
Locations (1):
- University of Oulu, Oulu, Finland

REFERENCES:
- [Background] Ahola R, Pyky R, Jamsa T, Mantysaari M, Koskimaki H, Ikaheimo TM, Huotari ML, Roning J, Heikkinen HI, Korpelainen R. Gamified physical activation of young men--a Multidisciplinary Population-Based Randomized Controlled Trial (MOPO study). BMC Public Health. 2013 Jan 14;13:32. doi: 10.1186/1471-2458-13-32. PMID 23311678
- [Derived] Leinonen AM, Pyky R, Ahola R, Kangas M, Siirtola P, Luoto T, Enwald H, Ikaheimo TM, Roning J, Keinanen-Kiukaanniemi S, Mantysaari M, Korpelainen R, Jamsa T. Feasibility of Gamified Mobile Service Aimed at Physical Activation in Young Men: Population-Based Randomized Controlled Study (MOPO). JMIR Mhealth Uhealth. 2017 Oct 10;5(10):e146. doi: 10.2196/mhealth.6675. PMID 29017991
- [Derived] Jauho AM, Pyky R, Ahola R, Kangas M, Virtanen P, Korpelainen R, Jamsa T. Effect of wrist-worn activity monitor feedback on physical activity behavior: A randomized controlled trial in Finnish young men. Prev Med Rep. 2015 Jul 22;2:628-34. doi: 10.1016/j.pmedr.2015.07.005. eCollection 2015. PMID 26844128